CLINICAL TRIAL: NCT01777464
Title: Role of the Central Nervous System in Allergic Rhinitis: Activation of Different Brain Regions After a Nasal Histamine Provocation in Healthy and Allergic Patients
Brief Title: Role of the Central Nervous System in Allergic Rhinitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: analysing images ongoing
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: september2012
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2014-09

CONDITIONS: House Dust Mite Allergy
MeSH Terms: conditions — Dust Mite Allergy | interventions — Histamine; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Experimental): patients allergic to house dust mite receive sham solution for 5 minutes on first visit and histamine (16mg/ml) for 5 minutes on second visit
  Interventions: Biological: histamine; Biological: sham
- healthy controls (Sham Comparator): healthy controls receive sham solution for 5 minutes on first visit and histamine (16mg/ml) for 5 minutes on second visit
  Interventions: Biological: histamine; Biological: sham

INTERVENTIONS:
Biological: histamine — administration of histamine solution (16 mg/ml) via aerosol for 5 minutes while lying under a fMRI scan
Biological: sham — sham solution

SUMMARY:
In order to evaluate the effects a nasal provocation on the activation of different brain regions, the investigators want to set up a clinical trial investigating the short-term effects of a nasal histamine provocation in healthy volunteers and allergic patients while in supine position under the functional MRI device in order to visualize different brain regions.

DETAILED DESCRIPTION:
Evaluate the effects a nasal provocation on the activation of different brain regions

ELIGIBILITY:
Inclusion Criteria:

* Patients with a positive skin prick test to grass pollen and with pollen allergic symptoms during the pollen season OR patients with a negative skin prick test and with no allergic symptoms during the pollen season.
* Age > 18 and < 50 years
* Written informed consent
* Willingness to adhere to visit schedules
* Adequate contraceptive precautions in female patients with childbearing potential

Exclusion Criteria:

* Current or recent (finished less than 2 years) immunotherapy against grass pollen.
* Systemic steroid treatment less than 6 weeks before the inclusion in the study.
* Nasal steroid spray, oral leukotriene antagonists or long-acting antihistamines less than 4 weeks before the inclusion.
* Presence of purulent secretions in nasal cavity.
* Severe septal deviation (septum reaching concha inferior or lateral nasal wall).
* Patient is pregnant or breastfeeding.
* Patient has any disorder of which the investigators feel at the time of evaluation for participation in the study that this may compromise the ability to give truly informed consent for participation in this study.
* Patient is currently enrolled in other investigational drug trial(s) or is receiving other investigational agent(s) for any other medical condition.
* No independent medication management in daily life or disability to perform fine motoric handling of medication
* Patients with asthma will be excluded.
* Patients suffering from claustrophobia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-11; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
brain activation | 5 minutes
  The specific aim of this study is to visualize the type and location of brain activation in healthy and allergic volunteers by a nasal provocation with histamine, using the functional MRI technology.

SECONDARY OUTCOMES:
nasal symptoms and Peak Nasal Inspiratory Flow | before and after scans
  Evaluation of nasal symptoms (runny nose, blocked nose, itchy nose and post-nasal drip) and conjunctival symptoms (lacrimation and itchy eyes) will be done with VAS scores and the Peak Nasal Inspiratory Flow (PNIF) will be measured before and after both functional MRI (fMRI) scans

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hellings, Dr, Principal Investigator — KU Leuven
Locations (1):
- uz leuven ORL, Leuven, Vlaams Brabant, Belgium